CLINICAL TRIAL: NCT02767648
Title: Inter-regional Cohort of Neonatal and Infant Cholestasis in the Greater Southwest Region
Acronym: CHOLESTASE
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 08 030 08; 2008 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2015-07-10; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Cholestasis
Keywords: cholestasis; neonatal; infant
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — proteomic urine analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cholestasis: infant suffering from cholestasis proteomic urine analysis
  Interventions: Other: proteomic urine analysis

INTERVENTIONS:
Other: proteomic urine analysis — proteomic urine analysis

SUMMARY:
The goal of the study is to characterize the epidemiologic data of the neonatal and infant cholestasis.

ELIGIBILITY:
Inclusion Criteria:

* Infant <1 year suffering from cholestasis

Exclusion Criteria:

* Rejection or inability for parent to give their informed consent

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infant suffering from cholestasis
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Gathering mother epidemiologic characteristics as assessed by pregancy informations collection | Day 1 (inclusion)
  Date of child birth, course of pregnancy, occurrence of twin pregnancy, serology abnormalities, family background of liver desease, course of previous pregnancies
Gathering new born epidemiologic characteristics as assessed by birth informations collection | Day 1 (inclusion)
  Birth anamnesis, inclusion age, hepatic desease history, hemostasis workup, validated etiologic diagnosis and criteria for the diagnosis, specific and non-specific therapeutic care
Epidemiologic characteristics follow up as assessed by medical monitoring | When children are between 12 and 18 months old
  Desease evolution in the first year of life, clinical evaluation, biological evaluation, final diagnosis, complications of the sickness, existence of transplatation, death

SECONDARY OUTCOMES:
Homogenization of diagnosis and treatment of new born with the constitution and follow up of a prospective cohorte | Up to 3 years
  Homogenize the care pathway of neonatal and infant cholestasis
Extend the study to the national french territory using the hepatology association network | Up to 3 years
  Use this study to start a national study
Identification of proteomic profiles using the biologic collection gathered in the cohorte population | Up to 3 years
  Identify one or more specific proteomic profile of neonatal cholestasis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Broue, MD, Principal Investigator — UH Toulouse; Thierry Lamireau, MD, Principal Investigator — University Hospital, Bordeaux; Jane Languepin, MD, Principal Investigator — UH Limoges; Sebastien Fournier-Favre, MD, Principal Investigator — UH Monptellier
Locations (4):
- France (4):
  - UH Bordeaux, Bordeaux
  - UH Limoges, Limoges
  - UH Montpellier, Montpellier
  - UH Toulouse, Toulouse